CLINICAL TRIAL: NCT06651086
Title: Hybrid Effectiveness-Implementation Trial of an Executive Functioning Intervention for Children's Mental Health Services
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, San Diego (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Kelsey Dickson, Associate Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS-2024-0105; R01MH137179 (NIH)
Record Dates: First submitted 2024-10-09; First posted 2024-10-21 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder; Executive Functioning
Keywords: Autism spectrum disorder; executive functioning; emotion regulation; mental health symptoms; Unified Protcol for Children; Unstuck and On Target; evidence based intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participating mental health programs from California and Colorado will be randomized to one of two conditions: Unstuck and On Target training and Unified Protocol for Children training. Therapists will be recruited from each participating program and enrolled as a dyad with target children. Autistic children will be enrolled at the beginning of therapist participation and before intervention training. Non-autistic children will be enrolled after intervention training and implementation or approximately 6 months after therapist enrollment. Participating therapists and child clients served in those programs will receive the same condition as their enrolled program.
Who Masked: Outcomes Assessor
Masking Description: Observational Coders Direct Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unstuck and On Target (Active Comparator): Unstuck and on Target (Unstuck; Cannon et al., 2021) is a cognitive-behavioral, intervention designed to be feasibly delivered by teachers and school staff in the elementary school setting. It was adapted for and pilot-tested in outpatient mental health. Unstuck targets key executive functions, including flexibility, goal-setting, planning, and coping. Sessions include prescribed content and activities to facilitate guided practice and home extension activities to aid generalization beyond the therapeutic session. It includes both child- and caregiver-directed strategies. It has been shown effective for youth with autism and attention-deficit/hyperactivity disorder.
  Interventions: Behavioral: Unstuck and On Target
- Unified Protocol for Children (Active Comparator): Unified Protocol for Children is a transdiagnostic, cognitive-behaviorally based treatment targeting shared core dysfunctions underlying emotional disorders, including distress intolerance and emotional dysregulation. It was developed by integrating cognitive-behavioral and mindfulness strategies and includes prescribed activities, in-vivo experiments, and home-extension components to promote generalization. It includes both child- and caregiver-directed strategies. In addition to its effectiveness for youth with emotional disorders, recent work supports its efficacy for youth with additional non-emotional disorders (e.g., externalizing challenges, irritability).
  Interventions: Behavioral: Unified Protocol for Children

INTERVENTIONS:
Behavioral: Unstuck and On Target — Unstuck and on Target (Unstuck; Cannon et al., 2021) is a cognitive-behavioral, intervention designed to be feasibly delivered by teachers and school staff in the elementary school setting. It was adapted for and pilot-tested in outpatient mental health. Unstuck targets key executive functions, including flexibility, goal-setting, planning, and coping. Sessions include prescribed content and activities to facilitate guided practice and home extension activities to aid generalization beyond the therapeutic session. It includes both child- and caregiver-directed strategies. It has been shown effective for youth with autism and attention-deficit/hyperactivity disorder.
  Arms: Unstuck and On Target
Behavioral: Unified Protocol for Children — Unified Protocol for Children is a transdiagnostic, cognitive-behaviorally based treatment targeting shared core dysfunctions underlying emotional disorders, including distress intolerance and emotional dysregulation. It was developed by integrating cognitive-behavioral and mindfulness strategies and includes prescribed activities, in-vivo experiments, and home-extension components to promote generalization. It includes both child- and caregiver-directed strategies. In addition to its effectiveness for youth with emotional disorders, recent work supports its efficacy for youth with additional non-emotional disorders (e.g., externalizing challenges, irritability).
  Arms: Unified Protocol for Children

SUMMARY:
This project aims to follow up on a prior project examining the impact of training therapists in an executive functioning intervention Unstuck and On Target (UOT) adapted for community mental health settings. Study aims are to test the clinical and implementation effectiveness of training mental health therapists in Unstuck and On Target, an executive functioning intervention, relative to Unified Protocol for Children, a transdiagnostic intervention for emotional disorders. This includes examining the implementation of Unstuck and associated outcomes (e.g., effective delivery, expanded use of Unstuck beyond autism, the feasibility of Unstuck) and impact on changes in child executive functioning and behaviors.

DETAILED DESCRIPTION:
Autism is a highly prevalent neurodevelopmental condition, affecting 1 in 36 youth. The annual cost in the U.S. of autism was $223 billion in 2020 and is estimated to rise to $589 billion by 2030. Outcomes are poor and care disparities and high rates of unmet service needs are common. Mental health services play a key role in caring for autistic youth. There have been efforts to develop evidence-based interventions (EBIs) with the potential to lessen the public health burden of autism. Yet, research indicates limited community EBI penetration. Several work gaps remain, including a focus on EBIs designed for community implementation and those addressing multilevel barriers impeding EBI use. There is an urgent need to focus on EBIs that improve mental health services for autism and optimize outcomes for this priority, complex population. Executive functioning (EF) is a potent mechanism underlying autism and commonly co-occurring mental health conditions. EF impairments (e.g., inflexibility, poor goal setting, poor planning) contribute to negative outcomes spanning multiple areas (e.g., academic, vocational, health). Our work underscores the impact of EF deficits on mental health services, including its transdiagnostic impact on the majority of children served in this setting and its role as a barrier to psychotherapy engagement and progress. EF is responsive to treatment, and mental health therapists cite a significant need and motivation for EF treatments, making EF EBIs highly relevant for community mental health settings. However, EF EBIs have not been widely used and tested in such settings. Autism EBIs, or those developed or adapted for autistic youth, have the potential to enhance mental health services, in addition to improving service quality for the populations targeted (e.g., autism). This is due to the specific components and strategies incorporated into the EBI to enhance its impact and fit. We propose a Hybrid Type 2 randomized trial examining the effectiveness and implementation of an autism EF EBI (Unstuck and On Target) in community mental health settings. Unstuck and On Target is a cognitive-behavioral EF intervention effective for autism.

With NIMH funding (K23MH115100;), Unstuck and On Target were systematically adapted for and tested in mental health settings, with a pilot test suggesting its preliminary effectiveness, high fidelity, and use beyond autism. Findings have the potential to transform implementation and service quality for the high-priority population of autistic youth as well as youth generally. Aim 1. Evaluate the effectiveness and implementation of an autism EBI (Unstuck and On Target), relative to a non-autism transdiagnostic intervention (Unified Protocol for Children) for autistic youth. Aim 2. Evaluate mediators of EBI training effects to confirm engaged change mechanisms of clinical and implementation outcomes. Aim 3. Explore the generalized effects of EBI training on reach and improved psychotherapy quality with non-autistic youth.

ELIGIBILITY:
Inclusion Criteria:

Mental Health Programs:

* Publicly-funded
* Providing outpatient or school-based psychotherapy services to children
* Have at least 8 mental health providers on staff

Therapists:

* Employed as staff or trainee at a participating program
* Employed at the program for at least the next 12 months
* Providing psychotherapy services to children
* Has an eligible child on current caseload (see below)

Autistic Child/Caregiver Participants (enrolled in a dyad with a participating therapist):

* Child age 6-12 years
* Receiving services from an enrolled therapist
* Documented or suspected* autism diagnosis

  * In the event of suspected autism diagnosis, the presence of elevated autism symptoms on the Social Responsiveness Scale-2nd Edition or the Autism Diagnostic Observation Scale-2nd Edition

Non-Autistic Child/Caregiver Participants (enrolled in a dyad with a participating therapist):

* Child age 6-12 years
* Receiving services from an enrolled provider
* No history of documented or suspected autism diagnosis

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 672 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Child Mental Health Symptoms | Pre-EBI implementation, 6-months post-EBI implementation, 12-month follow-up after EBI implementation
  Changes in mental health symptoms will be measured by the Child Behavior Checklist (CBCL), a 113-item rating scale measuring a range of mental health symptoms.
Externalizing Behaviors | Pre-EBI implementation, 6-months post-EBI implementation, 12-month follow-up after EBI implementation
  Primary outcome measures include externalizing behaviors. The Eyberg Child Behavior Inventory (ECBI), a 36-item widely used rating scale, will measure these behaviors.
Evidence-based Intervention Fidelity | During 6-month EBI implementation
  A trained observer masked to evidence-based intervention (EBI) condition and time will assess EBI delivery during recorded sessions of participating therapist-client dyads. Unique fidelity forms with items corresponding to each EBI (Unstuck and On Target and Unified Protocol for Children) will be used. Items rate adherence (i.e., the degree to which key components are delivered as intended) and competence (responsiveness, engagement, skill). Items are rated on a 1-5 scale, with higher scores indicating better fidelity. Measures have internal consistencies and are shown to be sensitive to treatment effects.
Evidence-Based Intervention Training Engagement | 6-months post-EBI implementation
  Therapist evidence-based intervention (EBI) training engagement will be operationalized as adherence to training requirements, including participation in training/consultation (as rated by trainers) and training-related submissions (forms, materials).

SECONDARY OUTCOMES:
Evidence-Based Intervention Reach | 6-months post-EBI implementation, 12-month follow-up after EBI implementation, 18-month follow-up after EBI implementation
  Therapists will report on evidence-based intervention (EBI) reach as operationalized by the number and types of clients (e.g., presenting problem, diagnostic profile) of clients treated with EBI, including specific components used. Measure was adapted from prior work and used in the PI's feasibility trial.
Psychotherapy Quality | 6-months post-EBI implementation
  Therapists will complete the Evidence-Based Practice Concordant Care Assessment-Therapist Report (ECCA). With funding from NIMH (R01MH100134; PI: Brookman-Frazee/Lau), ECCA was developed and validated as a pragmatic measure of evidence-based strategy delivery in psychotherapy sessions useful in indexing mental health quality of care. It has internal consistency and inter-rater reliability. Therapists will complete weekly regarding strategies within a given session with a participating client.

OTHER OUTCOMES:
Clinical Mediator: Changes in Executive Functioning, BRIEF-II | Pre-EBI implementation, 6-months post-EBI implementation, 12-month follow-up after EBI implementation
  Changes in executive functioning will be examined using several measures of executive functioning, including the Brief Rating Inventory of Executive Function-2nd Edition (BRIEF-II)- Parent Report, a 63-item rating scale supported by RDoC Working Group that measures real-world EF skills. This measure was shown to be sensitive to change in prior Unstuck trials, including PI's feasibility trial.
Clinical Mediator: Changes in Executive Functioning, EFCT | Pre-EBI implementation, 6-months post-EBI implementation, 12-month follow-up after EBI implementation
  Changes in executive functioning will be examined using several measures of executive functioning, including the Executive Function Challenge Task (EFCT), a standardized, semi-structured assessment of real-world EF abilities. This measure was shown to be sensitive to change in prior Unstuck trials, including PI's feasibility trial.
Clinical Mediator: Changes in Executive Functioning, DCCS | Pre-EBI implementation, 6-months post-EBI implementation, 12-month follow-up after EBI implementation
  Changes in executive functioning will be examined using several measures of executive functioning, including the NIH toolbox Dimensional Change Card Sort test (DCCS), a standard, lab-based task for assessing cognitive flexibility. This measure was shown to be sensitive to change in prior Unstuck trials, including PI's feasibility trial.
Clinical Mediator: Changes in Emotion Regulation | Pre-EBI implementation, 6-months post-EBI training, 12-month follow-up after EBI implementation
  Changes in Emotion Regulation will be examined using the Emotion Dysregulation Inventory (EDI), a 30-item parent-report ratings scale measuring emotion regulation.
Implementation Mediator: Changes in Intervention Perceptions of Fit, PCIS | Pre-EBI implementation, 6-months post-EBI implementation
  Changes in perceptions of fit regarding the evidence-based intervention will be examined using the Perceived Characteristics of Intervention Scale (PCIS), a 20-item measure assessing perceptions towards an intervention, including compatibility or fit.
Implementation Mediator: Changes in Intervention Perceptions of Fit, IAM | Pre-EBI implementation, 6-months post-EBI implementation
  Changes in perceptions of fit regarding the evidence-based intervention will be examined using the Intervention Appropriateness Measure (IAM), a 4-item measure that assesses the appropriateness or fit of an intervention.
Implementation Mediator: Changes in Autism Self-Efficacy and Knowledge, Confidence | Pre-EBI implementation, 6-months post-EBI implementation
  Changes in therapist autism self-efficacy and knowledge will be examined using the Therapist Confidence Scale for Autism Spectrum Disorder (TCS-ASD), a 14-item measure assessing confidence in psychotherapy for autistic clients.
Implementation Mediator: Changes in Autism Self-Efficacy and Knowledge, Knowledge | Pre-EBI implementation, 6-months post-EBI implementation
  Changes in therapist autism self-efficacy and knowledge will be examined using the Therapist Knowledge for Autistic Clients, a 6-item measure of knowledge of mental health-related topics for autism (e.g., core symptoms, co-occurring problems).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Diego State University, San Diego, California
  - University of Colorado - Anschutz, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Deidentitifed data will be shared with NDA
Supporting Information: Study Protocol
Time Frame: Will be reported per NDA timeline.
Access Criteria: Request login access to NDA

REFERENCES:
- [Background] Dickson KS, Galligan M, Holt T, Kenworthy L, Anthony L, Roesch S, Brookman-Frazee L. Randomized Feasibility Pilot of an Executive Functioning Intervention Adapted for Children's Mental Health Settings. J Autism Dev Disord. 2025 Jul;55(7):2407-2421. doi: 10.1007/s10803-024-06365-8. Epub 2024 Apr 28. PMID 38678517
- [Background] Dickson KS, Aarons GA, Anthony LG, Kenworthy L, Crandal BR, Williams K, Brookman-Frazee L. Adaption and pilot implementation of an autism executive functioning intervention in children's mental health services: a mixed-methods study protocol. Pilot Feasibility Stud. 2020 Apr 27;6:55. doi: 10.1186/s40814-020-00593-2. eCollection 2020. PMID 32699642
- [Derived] Dickson KS, Kennedy SM, Safer J, Brookman-Frazee L, Roesch S, Anthony LG. Study protocol for a hybrid type 2 effectiveness-implementation trial of two interventions for autistic and non-autistic youth in children's mental health settings: one tailored for neurodivergence and one universal. Implement Sci Commun. 2025 Nov 26;6(1):131. doi: 10.1186/s43058-025-00799-6. PMID 41299783